CLINICAL TRIAL: NCT01615692
Title: The Extension to Follow up Study of the Compression Stockings to Prevent the Post-Thrombotic Syndrome (SOX Trial)
Brief Title: The 36-month Extension to Follow up Sub Study
Status: Withdrawn | Type: Observational
Why Stopped: Sub study was not pursued as overall trial was negative
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Sigvaris Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Susan Kahn, SOX Trial Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: MOP-102610; ISRCTN71334751; NCT00143598 (Registry Identifier: ISRCTN; Clinicaltrials.gov)
Record Dates: First submitted 2012-06-01; First posted 2012-06-11 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Postphlebitic Syndrome; Post-Thrombotic Syndrome; Deep Vein Thrombosis
Keywords: Elastic Stockings; Stockings, Compression; Randomized Controlled Trials; Quality of Life
MeSH Terms: conditions — Postphlebitic Syndrome; Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 36-mth follow up visit: The cohort will consist of original subjects of the SOX Trial who consent to participate in the extension to follow up sub study.

SUMMARY:
The purpose of this study is to evaluate leg health for one additional year in patients with symptomatic proximal deep venous thrombosis who did not already develop Post-Thrombotic Syndrome (PTS) during the 2 years of follow up in the SOX Trial.

DETAILED DESCRIPTION:
The post-thrombotic syndrome (PTS) is a frequent, burdensome and costly condition that occurs in about one third of patients after an episode of deep vein thrombosis (DVT). Affected patients have chronic leg pain and swelling, and sometimes develop skin ulcers. At present, there is little to offer for the treatment of this condition. Prevention of PTS is the key to reducing its burden on patients and society. Elastic compression stockings (ECS) for two years following DVT could be helpful in preventing or delaying onset of PTS at three years, however data supporting this is limited.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a first, symptomatic, objectively confirmed proximal DVT diagnosed within the last 14 days (with or without concurrent distal DVT or pulmonary embolism)
* Who have no contraindications to standard treatment with heparin and/or warfarin, and
* Who provide informed consent to participate

Exclusion Criteria:

* Contraindication to compression stockings
* Limited lifespan (estimated < 6 months)
* Geographic inaccessibility preventing return for follow-up visits
* Inability to apply stockings daily and unavailability of a caregiver to apply stockings daily
* Treatment of acute DVT with thrombolytic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously enrolled in the SOX Trial (ClinicalTrials.gov Identifier NCT00143598) who did not develop PTS by 2 years follow up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of PTS and PTS severity | 3 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Susan R. Kahn, M.D., M.Sc., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (20):
- Canada (20):
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences - Chedoke Division, Hamilton, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences - Henderson General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre-Dame, Montreal, Quebec
  - Royal Victoria Hospital - McGill University Health Centre, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Centre, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec, Hôpital de l'Enfant-Jésus, Québec, Quebec

REFERENCES:
- [Background] Kahn SR, Shbaklo H, Shapiro S, Wells PS, Kovacs MJ, Rodger MA, Anderson DR, Ginsberg JS, Johri M, Tagalakis V; SOX Trial Investigators. Effectiveness of compression stockings to prevent the post-thrombotic syndrome (the SOX Trial and Bio-SOX biomarker substudy): a randomized controlled trial. BMC Cardiovasc Disord. 2007 Jul 24;7:21. doi: 10.1186/1471-2261-7-21. PMID 17711595